CLINICAL TRIAL: NCT06026943
Title: A Feasibility and Safety Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Locally Advanced Pancreatic Cancer
Brief Title: Alpha Radiation Emitters Device for the Treatment of Pancreatic Cancer Emitters for the Treatment of Locally Advanced Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PANC-03
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Unresectable Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; Unresectable Pancreatic Cancer; Pancreatic Adenocarcinoma; Alpha radiation; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: DaRT seeds insertion

INTERVENTIONS:
Device: DaRT seeds insertion — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms
  Other Names: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for advanced pancreatic cancer

DETAILED DESCRIPTION:
This is a prospective, interventional, single-center, open label, single arm study. The study is designed to evaluate the feasibility and Safety of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Locally Advanced Pancreatic Cancer

The study will be comprised of a screening period, DaRT insertion visit, 3 months follow up per subject and 2 years for accrual and trial completion. The total duration of the study will be 24 months from the DaRT insertion procedure.

15 patients with a safety interim analysis after the 5 first patients . patients with advanced pancreatic cancer will be recruited by the investigational site.

Eligible patients who meet inclusion/exclusion criteria (as assessed during the screening period) will be invited to the site for the procedure of DaRT seeds insertion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven NCCN locally advanced PC
* Patients must have i) received at least one line of chemotherapy (any kind) OR ii) are medically unfit for further chemotherapy, AND iii) the tumor is still not deemed as resectable with radical surgery, or the patient does not wish to go through surgery.
* DaRT indication validated by a multidisciplinary team.
* Measurable lesion per RECIST (version 1.1) criteria
* TC at Verona's center (not been over a month)
* Lesion size ≤ 5 cm in the longest diameter
* Age ≥18 years old
* ECOG Performance Status Scale ≤ 2
* Life expectancy is more than 6 months
* WBC ≥ 3500/μl, granulocyte ≥ 1500/μl
* Platelet count ≥60,000/μl
* Calculated or measured creatinine clearance ≥ 30cc/min. Calculated or measured creatinine clearance can be ≥ 40cc/min given stability of creatinine levels over the past three weeks (at least 1 test per week).
* AST and ALT ≤ 2.5 X upper limit of normal (ULN)
* INR < 1.4 for patients not on Warfarin
* Subjects are willing and able to sign an informed consent form
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after brachytherapy.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.

Exclusion Criteria:

* Concomitant chemotherapy or immunotherapy within the past 4 weeks
* Prior radiation therapy to the pancreas
* CA 19-9 > 1000 Units/ml
* Fit for surgical exploration unless the patient refuses surgery
* Known hypersensitivity to any of the components of the treatment.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy (not including cholangitis) or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
* Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Breastfeeding women or women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 3 months after RT.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility- DaRT seed placement | Immediately following the insertion procedure
  Feasibility will be determined according to the rate of successful placement of DaRT seeds via imaging
Safety- Adverse events, Safety will be determined according to the overall incidence of device-related SAE's graded according to CTCAE v5.0 criteria | from DaRT-insertion up to 48 hours
  Safety will be determined according to the overall incidence of device-related SAE's graded according to CTCAE v5.0 criteria

SECONDARY OUTCOMES:
To evaluate the Efficacy of the Alpha DaRT seeds for locally advanced pancreatic cancer | 1 months and 3 months
  Local control evaluation according to RECIST v1.1
To evaluate the Efficacy of the Alpha DaRT seeds by measuring the CA-19-9 markers levels | 1 months and 3 months
  Change in CA 19-9 levels
Efficacy - to evaluate what is the percent of the Tumor Coverage by the Alpha DaRT seeds | immediately following the insertion procedure]
  Tumor Coverage
Efficacy- Alpha DaRT seeds | from DaRT-insertion up to initiation of a possible postablation therapy or up to a maximum three months
  Overall incidence of device-related SAE's graded according to CTCAE v5.0 criteria

OTHER OUTCOMES:
Exploratory Objective -to evaluate the changes in the immune markers by Blood samples for immune response | 1 month
  Changes in immune markers following treatment ,These biomarkers include:
  * CD3
  * CD4
  * CD8
  * CD69
  * CD137

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Paiella, MD, Principal Investigator — Pancreas Institute - Integrated University Hospital of Verona
Locations (1):
- Chirurgia Generale e del Pancreas, Istituto del Pancreas, Verona, Italy